CLINICAL TRIAL: NCT01714323
Title: Comparative Effectiveness of Post-Discharge Strategies for Hospitalized Smokers
Acronym: Helping HAND2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pittsburgh (Other); North Shore Medical Center (Other)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL111821 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder
Keywords: Cigarette smoking; Tobacco smoking; Tobacco use disorder
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Other): At discharge, the participant receives the standard care provided by the hospital. This consists of a handout with information to contact the state telephone quitline for additional smoking cessation support and to use smoking cessation medication as recommended by the hospital smoking counselor.
  Interventions: Behavioral: Standard Care
- Sustained Care (Experimental): A 3-month program after hospital discharge with these 2 components: (1) Free Medication and (2) Interactive Voice Response (IVR) Triage to Telephone Counseling.
  Interventions: Behavioral: Sustained Care

INTERVENTIONS:
Behavioral: Sustained Care — A 3-month program after hospital discharge with these 2 components: (1) Free Medication - A 30-day supply of FDA-approved medication (nicotine replacement, bupropion, or varenicline) given at hospital discharge and refillable for a total of 90 days to encourage medication use and adherence; (2) Interactive Voice Response (IVR) Triage to Telephone Counseling from a national quitline provider (Alere Wellbeing, Inc., previously Free & Clear). IVR aims to encourage medication adherence and enhance counseling efficiency by identifying smokers who need post-discharge support. Immediate transfer of a patient from automated IVR call to live telephone counselor will facilitate a successful connection to counseling.
  Arms: Sustained Care
Behavioral: Standard Care — Standard care consists of a handout with information about how to contact the state telephone quitline for additional smoking cessation support and to use smoking cessation medication as recommended by the hospital smoking counselor.
  Arms: Standard care

SUMMARY:
Cigarette smoking is the leading preventable cause of death in the U.S. The 2008 US Public Health Service Smoking Cessation Guideline recommends offering effective treatment to smokers in all health care settings, including hospitals. Nearly 4 million smokers are hospitalized each year, and hospital admission offers a "teachable moment" for intervention. Hospital-initiated smoking cessation intervention is effective, but only if contact continues for more than 1 month after discharge. The challenge is to translate this research into clinical practice by identifying an evidence-based cost-effective model that U.S. hospitals can adopt. The major barrier is sustaining contact after discharge. This project tests an innovative strategy to streamline the delivery and maximize the uptake of post-discharge smoking interventions.

Specific Aim: To test the effectiveness of an innovative strategy to maximize smokers' use of evidence-based tobacco treatment (counseling and medication) after hospital discharge, thereby increasing the proportion of smokers who achieve long-term (6-month) tobacco abstinence.

Study Design: A multi-site randomized controlled comparative effectiveness trial will enroll 1350 adult smokers admitted to 3 acute care hospitals in Massachusetts and Pennsylvania. All subjects will receive a brief in-hospital smoking intervention and be randomly assigned at discharge to either Standard Care (passive referral to their state quitline) or Extended Care, a 3-month program consisting of (1) Free Medication: A 30-day supply of FDA-approved medication (nicotine replacement, bupropion, or varenicline) given at hospital discharge and refillable for a total of 90 days to encourage medication use and adherence; (2) Interactive Voice Response (IVR) Triage to Telephone Counseling from a national quitline provider. IVR aims to encourage medication adherence and enhance counseling efficiency by identifying smokers who need post-discharge support. Immediate transfer of a patient from automated IVR call to live telephone counselor will facilitate a successful connection to counseling.

Outcomes, assessed at 1, 3, and 6 months after hospital discharge, are: (1) intervention effectiveness (cotinine-validated 7-day point-prevalence tobacco abstinence rate at 6 month follow-up [primary outcome] and other tobacco abstinence measures); (2) treatment utilization, and (3) cost-effectiveness (cost per quit). Exploratory analyses will examine the intervention's effect on hospital readmissions and mortality in the 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smoker (smoked at least 1 cigarette in the month before hospital admission and at least 1 cigarette per day when smoking at baseline rate in the month before hospital admission)
* Counseled by hospital smoking counselor during hospital stay
* Plans to stop smoking tobacco products after hospital discharge
* Agrees to take home a supply of smoking cessation medication after discharge
* Agrees to and able to accept telephone calls after hospital discharge

Exclusion Criteria:

* No access to a telephone or unable to communicate by telephone
* Severe psychiatric or neurologic disease precluding ability to provide informed consent and to be counseled
* Pregnant, nursing, or planning to become pregnant in next 3 months
* Unable to speak English
* Medical instability precluding study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1359 (Actual)
Dates: Start 2012-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Triant VA, Grossman E, Rigotti NA, Ramachandran R, Regan S, Sherman SE, Richter KP, Tindle HA, Harrington KF. Impact of Smoking Cessation Interventions Initiated During Hospitalization Among HIV-Infected Smokers. Nicotine Tob Res. 2020 Jun 12;22(7):1170-1177. doi: 10.1093/ntr/ntz168. PMID 31687769
- [Derived] Streck JM, Chang Y, Tindle HA, Regan S, Park ER, Levy DE, Singer DE, Ylioja T, Rigotti NA. Smoking Cessation After Hospital Discharge: Factors Associated With Abstinence. J Hosp Med. 2018 Nov 1;13(11):774-778. doi: 10.12788/jhm.2997. Epub 2018 Aug 29. PMID 30156578
- [Derived] Rigotti NA, Chang Y, Tindle HA, Kalkhoran SM, Levy DE, Regan S, Kelley JHK, Davis EM, Singer DE. Association of E-Cigarette Use With Smoking Cessation Among Smokers Who Plan to Quit After a Hospitalization: A Prospective Study. Ann Intern Med. 2018 May 1;168(9):613-620. doi: 10.7326/M17-2048. Epub 2018 Mar 27. PMID 29582077
- [Derived] Rigotti NA, Chang Y, Rosenfeld LC, Japuntich SJ, Park ER, Tindle HA, Levy DE, Reid ZZ, Streck J, Gomperts T, Kelley JHK, Singer DE. Interactive Voice Response Calls to Promote Smoking Cessation after Hospital Discharge: Pooled Analysis of Two Randomized Clinical Trials. J Gen Intern Med. 2017 Sep;32(9):1005-1013. doi: 10.1007/s11606-017-4085-z. Epub 2017 Jun 14. PMID 28616847
- [Derived] Rigotti NA, Tindle HA, Regan S, Levy DE, Chang Y, Carpenter KM, Park ER, Kelley JH, Streck JM, Reid ZZ, Ylioja T, Reyen M, Singer DE. A Post-Discharge Smoking-Cessation Intervention for Hospital Patients: Helping Hand 2 Randomized Clinical Trial. Am J Prev Med. 2016 Oct;51(4):597-608. doi: 10.1016/j.amepre.2016.04.005. PMID 27647060
- [Derived] Reid ZZ, Regan S, Kelley JH, Streck JM, Ylioja T, Tindle HA, Chang Y, Levy DE, Park ER, Singer DE, Carpenter KM, Reyen M, Rigotti NA. Comparative Effectiveness of Post-Discharge Strategies for Hospitalized Smokers: study protocol for the Helping HAND 2 randomized controlled trial. BMC Public Health. 2015 Feb 7;15:109. doi: 10.1186/s12889-015-1484-0. PMID 25879193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of eligible daily smokers admitted to 3 hospitals (Massachusetts General Hospital, Boston, MA; University of Pittsburgh Medical Center, Pittsburgh, PA; and North Shore Medical Center, Salem, MA) occurred during the period 12/3/2012 - 7/18/2014
Pre-assignment Details: 1359 patients were enrolled in the study and randomized to Sustained Care (n=681) or Standard Care (n=678). Two patients, 1 in each group, were excluded post-randomization but before hospital discharge (when intervention began) because they were not eligible. ITT analysis was conducted on 1357 patients (Standard Care n=677, Sustained Care n=680).
Period: Overall Study
Arm/Group | Standard Care | Sustained Care
Started | 677 | 680
Completed | 513 | 508
Not Completed | 164 | 172

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Sustained Care | Total
Number analyzed (Participants) | 677 | 680 | 1357
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.4) | 49.6 (12.8) | 49.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336 | 332 | 668
  Male | 341 | 348 | 689
Region of Enrollment [Number; unit: participants]
  United States | 677 | 680 | 1357

OUTCOME MEASURES:

1. Primary Outcome: Tobacco Abstinence - 6 Month Follow-up
Description: Cotinine-validated 7-day point prevalence tobacco abstinence at 6 month follow-up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
Participants | 105 | 113
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; Data from all three sites were combined after determining that outcomes did not vary by hospital using Breslow-Day tests. The proportion abstinent by treatment arm was assessed using chi-square test; Test type: Superiority or Other; p > 0.05, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.84 to 1.37]

2. Secondary Outcome: Continuous Tobacco Abstinence
Description: Continuous tobacco abstinence after hospital discharge assessed by self-report at 1, 3, and 6 months.
Time Frame: 1 month, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
Participants
  1 month follow-up | 179 | 211
  3 month follow-up | 122 | 147
  6 month follow-up | 101 | 121
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Point Prevalence Tobacco Abstinence
Description: 7-day point prevalence tobacco abstinence after hospital discharge, assessed by self-report
Time Frame: 1 month, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
Participants
  1 month follow-up | 217 | 295
  3 month follow-up | 206 | 253
  6 month follow-up | 180 | 209
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; This compares at Month 1; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Standard Care vs Sustained Care; This is analysis for Month 3; Test type: Superiority; p < 0.01, Chi-squared
Statistical Analysis 3: Comparison: Standard Care vs Sustained Care; This is for Month 6; Test type: Superiority; p < 0.09, Chi-squared

4. Secondary Outcome: Duration of Tobacco Abstinence After Hospital Discharge
Description: Self-reported number of days in which a participant was abstinent from tobacco after hospital discharge, by self-report, obtained from surveys done at 1 month, 3 months, and 6 months. Patient can only relapse once but it can occur at any point up to 6 months after discharge. Therefore, the data point can come from either the 1 or 3 or 6 month follow-up depending on when relapse occurred.
Time Frame: 1 month, 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
days | 7 [2 to 75] | 14 [3 to 90]

5. Secondary Outcome: Use of Smoking Cessation Treatment After Hospital Discharge
Description: Use of either FDA-approved pharmacotherapy for tobacco dependence (nicotine replacement therapy, bupropion, or varenicline), or psychosocial support (including telephone counseling, in person counseling, web-based counseling, physician counseling).
Time Frame: 1 month, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
Participants
  1 month follow-up | 306 | 491
  3 month follow-up | 404 | 554
  6 month follow-up | 448 | 580
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; Test type: Superiority or Other; p < 0.001, Chi-squared — This is the p value for the comparison at each follow up point: 1 mo, 3 mo, and 6 mo

6. Other Pre Specified Outcome: All-cause Hospitalizations
Description: Self-reported admission to a hospital in the 12 months after the index hospitalization.
Time Frame: 12 months
Measure: Number; unit: hospital admissions
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
hospital admissions | 224 | 216
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; Test type: Superiority or Other; p > 0.05, Chi-squared

7. Other Pre Specified Outcome: All-cause Mortality
Description: Death from any cause in the 6 months after hospital discharge
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Sustained Care
Number analyzed (Participants) | 677 | 680
Participants | 14 | 13
Statistical Analysis 1: Comparison: Standard Care vs Sustained Care; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year (hospital readmissions); 6 months (deaths)
Description: Hospital admissions for 1 year after index hospitalization were obtained by chart review of admissions to the network of hospitals affiliated with Partners HealthCare and University of Pittsburgh Medical Center. Deaths in the first 6 months were systematically identified at patient assessments (1, 3, and 6 months). No systematic assessment of other adverse events during the trial was done due to the intervention's minimal risk.
Arm/Group | Standard Care | Sustained Care
Serious Adverse Events (participants affected / at risk) | 224/677 | 216/680
Other Adverse Events (participants affected / at risk) | 0/677 | 0/680
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care (N=677) | Sustained Care (N=680)
Hospital Readmission (Gastrointestinal disorders) | 66 | 70
Hospital Readmission (Blood and lymphatic system disorders) | 19 | 4
Hospital Readmission (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Hospital Readmission (Cardiac disorders) | 50 | 48
Hospital Readmission (Skin and subcutaneous tissue disorders) | 21 | 15
Hospital Readmission (Endocrine disorders) | 10 | 25
Hospital Readmission (Eye disorders) | 2 | 1
Hospital Readmission (General disorders) | 22 | 13
Hospital Readmission (Infections and infestations) | 15 | 7
Hospital Readmission (Injury, poisoning and procedural complications) | 44 | 31
Hospital Readmisson (Hepatobiliary disorders) | 20 | 22
Hospital Readmission (Metabolism and nutrition disorders) | 17 | 35
Hospital Readmission (Musculoskeletal and connective tissue disorders) | 15 | 8
Hospital Readmission (Nervous system disorders) | 9 | 17
Hospital Readmission (Psychiatric disorders) | 29 | 19
Hospital Readmission (Respiratory, thoracic and mediastinal disorders) | 26 | 29
Hospital Readmission (Vascular disorders) | 24 | 31
Death (Cardiac disorders) | 7 | 2
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Death (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (Hepatobiliary disorders) | 2 | 1
Death (Infections and infestations) | 2 | 4
Death (Injury, poisoning and procedural complications) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes